CLINICAL TRIAL: NCT05606445
Title: Understanding and Objectively Measuring Paratonia in Persons With Dementia: a Surface Electromyography Approach
Brief Title: Surface EMG to Measure Paratonia in Dementia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Hanzehogeschool Groningen (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL81562.042.22
Record Dates: First submitted 2022-09-27; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Dementia Alzheimers
Keywords: Paratonia; Neuromotor
MeSH Terms: conditions — Alzheimer Disease; Muscle Rigidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- 1: Healthy young (18-30 years old) (n = 40). This group will be used to assess the development of paratonia in healthy conditions.
  Interventions: Behavioral: Elbow movement
- 2: Healthy middle aged (40-55y) (n = 40). This group will be used to assess the development of paratonia in healthy conditions.
  Interventions: Behavioral: Elbow movement
- 3: Healthy old (>65y) (n = 40). This group will be used to assess the development of paratonia in healthy conditions.
  Interventions: Behavioral: Elbow movement
- 4: People with mild cognitive impairment (n = 40). This group will be used to assess the severity of paratonia in the various stages of dementia.
  Interventions: Behavioral: Elbow movement
- 5: People with mild dementia according to the Clinical Dementia Rating (n = 40). This group will be used to assess the severity of paratonia in the various stages of dementia.
  Interventions: Behavioral: Elbow movement
- 6: People with moderate dementia according to the Clinical Dementia Rating (n = 40). This group will be used to assess the severity of paratonia in the various stages of dementia.
  Interventions: Behavioral: Elbow movement
- 7: People with severe dementia according to the Clinical Dementia Rating (n = 40). This group will be used to assess the severity of paratonia in the various stages of dementia.
  Interventions: Behavioral: Elbow movement

INTERVENTIONS:
Behavioral: Elbow movement — The behavioral paradigm consist of a passive and active movement condition. Both conditions consist of arm movements along the entire range of motion by moving the distal segment of the arm towards the proximal segment and back under varying conditions. In the 'passive' condition, this arm movement will be performed by researcher at 3 different velocities in sinusoidal (continuous) and linear (non-continuous) fashions whereas in the 'active' condition, the participant will be instructed to move the arm in one velocity under internal and external focus of attention.

SUMMARY:
Rationale: A prominent and degenerative motor symptom of dementia is paratonia that heavily affects quality of life. However, paratonia is poorly recognized and the diagnosis yet relies on subjective evaluation by caregivers.

Objective: The primary aim of the proposed study is to develop a surface-electromyography-based method to objectively quantify paratonia in people with dementia. In addition, we aim to increase the understanding of the role of neuromuscular dysfunctions that contribute to paratonia.

Study design: Cross-sectional study, in people of various ages and at older age with different levels of cognitive impairment and neuromuscular functioning, in which we will examine the association between their physical and cognitive function and neuromuscular outcome measures.

Study population: Healthy young (18-30y, n = 40), middle-age (40-55y, n = 40) and older adults (>65y; n = 40). In addition, people with mild cognitive impairment (n = 40) as well as people with mild (n = 40), moderate (n = 40) and severe (n = 40) dementia.

Main study parameters/endpoints: Cognitive function, physical function, neuromuscular function expressed by muscle- and brain activity as well as coordination.

DETAILED DESCRIPTION:
Nearly 300.000 people in the Netherlands and approximately 55 million people worldwide (WHO) suffer from dementia. With 60 - 70% of all cases, Alzheimer's disease (AD) is the most common form of dementia. While AD is mostly associated with cognitive dysfunction, motor symptoms - as acknowledged in DSM-5 - are part of the neurocognitive domain and have shown to precede cognitive decline in people with AD. These data highlight that dementia not only involves cognitive but also motor components. As such, objective screening tools that can detect these motor symptoms are critical yet unavailable.

A prominent and degenerative motor symptom related to AD is paratonia. Paratonia was first described almost two centuries ago and defined as increased muscle tone during passive movements that is proportional to the strength of the stimulus applied up to the production of counter-movements in the later stages of dementia. Paratonia, therefore, is a motor symptom of AD that heavily affects the quality of life and is often misunderstood and mistaken for behavior of a psychosocial nature. However, despite their impact, motor symptoms of AD receive surprisingly little attention. Indirect evidence suggests that paratonia results from central, i.e., frontal lobe disinhibition, as well as peripheral, i.e., impaired skeletal muscle function due to collagen cross-linking and intramuscular inflammation. Based on these data, it can be argued that paratonia can be objectively quantified using non-invasive electrophysiological measurements. Once developed, such accessible and low-cost screening tool provide evidence for the presence and severity of motor symptoms of dementia in clinical settings besides symptoms of cognitive decline.

Currently, the presence and severity of paratonia are assessed with, respectively, the subjective paratonia assessment instrument (PAI) and the subjective Modified Ashworth Scale for Paratonia (MAS-P). However, objective tools to examine paratonia in people with dementia are not available and as such, the diagnosis of paratonia relies solely on subjective interpretation of clinicians. In a recent review, our research group highlighted the various gaps of knowledge in paratonia-research related to the poor recognition of paratonia and the lack of clear guidance for health professionals. Because eExperimental evidence suggested the possibility to measure paratonia through muscle activity. ,This possibility arises from the hypothesis that the increased muscle tone results from lesions in the frontal cortex in people with dementia and consequently increased disinhibition of the motor cortex. In addition, it is also possible that the heightened muscle tone is (partly) caused by disturbed interactions between ascending sensory inputs and descending motor output. As such, it is reasonable to hypothesize paratonia can be objectively characterized by neurophysiological motor and corticomotor parameters. Moreover, there are indications that motor symptoms precede cognitive decline in people with dementia. Therefore, the goals of the proposed project are threefold and focus on (1) examining whether it is possible to the development of an objectively and non-invasively quantifyassessment the development of paratonia with a tool method based on surface electromyography (sEMG) to quantify paratonia, (2) examining the development of the relationship between motor symptoms of AD and cognitive and physical function from preclinical healthy adults to increasing severity of dementia and (3) identifying the contribution of underlying neuromuscular dysfunctions that are associated with the development of paratonia.

ELIGIBILITY:
In order to be eligible to participate in this study, healthy participants must meet all of the following criteria:

* Age within one of the age-ranges described above.
* Intact cognitive function (MOCA > 26).

As for the people with AD, we will use the following inclusion criteria:

* Diagnosed mild cognitive impairment (CDR score 0.5), mild dementia (CDR score 1), moderate dementia (CDR score 2) or severe dementia (CDR score 2).
* Able to sit independently.

A potential healthy participant who meets any of the following criteria will be excluded from participation in this study:

* A history of central neurological problems (e.g. cerebral vascular attacks, epilepsy, acquired brain damage or Parkinson's Disease) or peripheral nerve problems.
* Intake of medication that substantially affects the functioning of the nervous system in the three months prior to the assessment. This includes psychotropic medication (ATC codes N03A, N05A, N05B, N05C, N06A, N06B), anti-migraine and analgesics.

A potential participant with dementia will be excluded from participation if:

* The participant has experienced intercurrent diseases that negatively affected cognitive and motor function.
* The participant has a fever at the time of the assessment.
* The participant is deliriant.
* The participant is terminally ill (i.e., life expectancy < 2 weeks according to the attending physician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We aim to include healthy young (18 - 30 y, n = 40), middle-aged (40 - 55 y, n = 40) and older adults (> 65 y; n = 40). In addition, we aim to include people with mild cognitive impairment (n = 40) as well as people with mild AD (n = 40), moderate AD (n = 40) and severe AD (n = 40). The severity of AD will be determined using the Clinical Dementia Rating.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Root mean square | The measure 'root mean square' will be computed from electromyography data acquired during the session on Day 1 of the experiment.
  From EMG data measured during flexion and extension movements, we will calculate the root mean square to assess the influence of movement velocity and shape as well as focus of attention on agonist and antagonist muscle activity.
Co-contraction index | The measure 'co-contraction index' will be computed from electromyography data acquired during the session on Day 1 of the experiment.
  From EMG data measured during flexion and extension movements, we will calculate the co-contraction index to assess the influence of movement velocity and shape as well as focus of attention on the control of agonist and antagonist muscle activity.
corticomuscular coherence | The measure 'corticomuscular coherence' will be computed from electromyography and electroencephalography data acquired during the session on Day 1 of the experiment.
  From EMG and EEG data measured during flexion and extension movements, we will calculate the corticomuscular coherence to assess the influence of movement velocity and shape as well as focus of attention on the connectivity between the brain and the muscles involved in the movement.
corticokinematic coherence | The measure 'corticokinematic coherence' will be computed from electroencephalography and goniometer data acquired during the session on Day 1 of the experiment.
  From goniometer and EEG data measured during flexion and extension movements, we will calculate the corticokinetic coherence to assess the influence of movement velocity and shape as well as focus of attention on the proprioceptive function during the involved movements.

SECONDARY OUTCOMES:
cognitive function | The measure 'cognitive function' will be estimated from the Montreal Cognitive Assessment taken on Day 1 of the experiment.
  As a measure of cognitive function, we will use the Montreal Cognitive Assessment.
physical function | The measure 'physical function' will be estimated from the Timed Up and Go test taken on Day 1 of the experiment.
  As a measure of physical function, we will use the Timed-Up and Go test and measure the time it takes (in seconds) to rise from a chair and walk three meters at comfortable speed, walk back and get seated again.

IPD SHARING:
Plan to Share IPD: No